CLINICAL TRIAL: NCT00900692
Title: Dynamic Splinting for Excessive Pronation Following CVA: A Randomized, Controlled Tial
Brief Title: Dynamic Splinting for Excessive Pronation Following CVA
Acronym: SupPro Botox
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009.001
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Pronation Contracture
Keywords: Excessive pronation; CVA; Forearm; Excessive pronation following CVA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynasplint Group (Experimental): Along with the standard of care Botox and manual therapy, patients will use the Supination Dynasplint every day
  Interventions: Device: Dynasplint
- Standard of care (No Intervention): Patients in the standard of care group will have the standard Botox treatments and manual therapy with no additional interventions.

INTERVENTIONS:
Device: Dynasplint — Dynamic splinting utilizes the protocols of Low-Load Prolonged Stretch (LLPS) with calibrated adjustable tension to increase Total End Range Time (TERT)to reduce contracture. The Dynasplint or "Experimental" group will add this therapy to their standard of care regimen
  Arms: Dynasplint Group

SUMMARY:
The purpose of this study is to examine range of motion and lasting effects of Botox injections along with the use of the Supination Dynasplint.

ELIGIBILITY:
Inclusion Criteria

Patients enrolled will have been diagnosed with excessive pronation following a stroke and will display the following symptoms:

* Pronation Contracture
* Ability to provide consent and follow directions as related to the protocol

Exclusion Criteria

* Treatment with Benzodiazepines
* Treatment with Baclofen (pump or oral)
* Treatment with Dantrolene sodium
* Treatment with Tizanidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
ROM changes with use of treatment | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Duerden, MD, Principal Investigator — Rehabilitation Associates of Indiana
Locations (1):
- Rehabilitation Associates of Indiana, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Andreasen DS, Aviles AA, Allen SK, Guthrie KB, Jennings BR, Sprigle SH. Exoskeleton for forearm pronation and supination rehabilitation. Conf Proc IEEE Eng Med Biol Soc. 2004;2004:2714-7. doi: 10.1109/IEMBS.2004.1403778. PMID 17270837
- [Background] Winchester P, McColl R, Querry R, Foreman N, Mosby J, Tansey K, Williamson J. Changes in supraspinal activation patterns following robotic locomotor therapy in motor-incomplete spinal cord injury. Neurorehabil Neural Repair. 2005 Dec;19(4):313-24. doi: 10.1177/1545968305281515. PMID 16263963
- [Background] Cooper. Et al. Proceedings of the Stroke Disparities Advisory Panel Meeting, Nov 08, 2002, Bethesda MD, National Institute of Neurological Disorders and Stroke
- [Background] McKinley W, Tewksbury MA, Sitter P, Reed J, Floyd S. Assistive technology and computer adaptations for individuals with spinal cord injury. NeuroRehabilitation. 2004;19(2):141-6. PMID 15201473
- [Background] Horsley SA, Herbert RD, Ada L. Four weeks of daily stretch has little or no effect on wrist contracture after stroke: a randomised controlled trial. Aust J Physiother. 2007;53(4):239-45. doi: 10.1016/s0004-9514(07)70004-1. PMID 18047458
- [Background] Nuismer BA, Ekes AM, Holm MB. The use of low-load prolonged stretch devices in rehabilitation programs in the Pacific northwest. Am J Occup Ther. 1997 Jul-Aug;51(7):538-43. doi: 10.5014/ajot.51.7.538. PMID 9242860
- [Background] Bloemen-Vrencken JH, de Witte LP, Post MW. Follow-up care for persons with spinal cord injury living in the community: a systematic review of interventions and their evaluation. Spinal Cord. 2005 Aug;43(8):462-75. doi: 10.1038/sj.sc.3101750. PMID 15838530
- [Background] Tsao CC, Mirbagheri MM. Upper limb impairments associated with spasticity in neurological disorders. J Neuroeng Rehabil. 2007 Nov 29;4:45. doi: 10.1186/1743-0003-4-45. PMID 18047660
- [Background] Bryden AM, Kilgore KL, Lind BB, Yu DT. Triceps denervation as a predictor of elbow flexion contractures in C5 and C6 tetraplegia. Arch Phys Med Rehabil. 2004 Nov;85(11):1880-5. doi: 10.1016/j.apmr.2004.01.042. PMID 15520985
- [Background] Lannin NA, Herbert RD. Is hand splinting effective for adults following stroke? A systematic review and methodologic critique of published research. Clin Rehabil. 2003 Dec;17(8):807-16. doi: 10.1191/0269215503cr682oa. PMID 14682551
- [Background] Naik AK, Pathirathna S, Jevtovic-Todorovic V. GABAA receptor modulation in dorsal root ganglia in vivo affects chronic pain after nerve injury. Neuroscience. 2008 Jul 17;154(4):1539-53. doi: 10.1016/j.neuroscience.2008.04.061. Epub 2008 May 3. PMID 18554816
- [Background] Mahmood NS, Kadavigere R, Avinash KR, Rao VR. Magnetic resonance imaging in acute cervical spinal cord injury: a correlative study on spinal cord changes and 1 month motor recovery. Spinal Cord. 2008 Dec;46(12):791-7. doi: 10.1038/sc.2008.55. Epub 2008 Jun 10. PMID 18542094
- [Background] Harvey L, de Jong I, Goehl G, Mardwedel S. Twelve weeks of nightly stretch does not reduce thumb web-space contractures in people with a neurological condition: a randomised controlled trial. Aust J Physiother. 2006;52(4):251-8. doi: 10.1016/s0004-9514(06)70004-6. PMID 17132119
- [Background] Patrick JH, Farmer SE, Bromwich W. Muscle stretching for treatment and prevention of contracture in people with spinal cord injury. Spinal Cord. 2002 Aug;40(8):421-2; author reply 423. doi: 10.1038/sj.sc.3101340. No abstract available. PMID 12124669
- [Background] Lai JM, Francisco GE, Willis FB. Dynamic splinting after treatment with botulinum toxin type-A: a randomized controlled pilot study. Adv Ther. 2009 Feb;26(2):241-8. doi: 10.1007/s12325-008-0139-2. Epub 2009 Feb 4. PMID 19194671